CLINICAL TRIAL: NCT00845585
Title: Ovine Graft (Omniflow II) Versus PTFE in Below Knee Arterial Reconstruction: A Prospective Randomized Multi Centre Study
Brief Title: Ovine Graft (Omniflow II) Versus PTFE in Below Knee Arterial Reconstruction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: found not enough centers for recruitment
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Jürg Schmidli, MD, Chief of Vascular Surgery, Dept of Cardiovascular Surgery, University Hospital Bern
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 114/08
Record Dates: First submitted 2009-02-16; First posted 2009-02-18 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2010-11

CONDITIONS: Peripheral Arterial Occlusive Disease
Keywords: arterial reconstruction; bypass; below knee; PZFE; Ovine graft; Omniflow II; graft patency
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Owniflow II (Active Comparator)
  Interventions: Device: Below Knee Arterial Reconstruction
- PTFE (Active Comparator)
  Interventions: Device: Below Knee Arterial Reconstruction

INTERVENTIONS:
Device: Below Knee Arterial Reconstruction — Patency, Reinterventions, Amputations, mortality
  Arms: Owniflow II
Device: Below Knee Arterial Reconstruction — Patency, Reinterventions, Amputations, mortality
  Arms: PTFE

SUMMARY:
The study intends to compare commonly used PTFE grafts with the biologic ovine graft Ominiflow II for below-knee bypass surgery in patients with peripheral artery occlusive disease with no autologous vein graft available. The hypothesis of this randomized trial is that that Omniflow II does not have a higher patency than PTFE over 36 months (one-sided test). An interim analysis will be performed at 18

DETAILED DESCRIPTION:
Background

Despite advances in endovascular therapies, arterial bypass to restore blood flow to a patent distal artery often is the best option in the management of lower extremity occlusive arterial disease. The greater saphenous vein is the conduit of choice for infrainguinal reconstructions - but it is not always available or is otherwise unusable in a significant percentage of patients. In those situations, arterial reconstruction using prosthetic material is an option. Synthetic and biological vascular grafts have been used for some three decades. With time, synthetic conduits tend to increase their thrombogenic potential rather than diminish it by formation of neointima. Over time biological grafts have become alternatives to synthetic materials, mainly in the more demanding applications below the knee. For various reasons most biological grafts have been withdrawn from the market and Omniflow II (Bio Nova International, Mel-bourne, Australia) is currently the only biological vascular prosthesis available for peripheral revascularisation.

Objective

The Omniflow II prosthesis is a biosynthetic device formed from stabilised sheep collagen with an integral polyester mesh. It is produced by inserting polyester mesh-covered mandrels beneath the cutaneous trunci muscle of adult sheep for a period of 12-14 weeks. The collagen-encapsulated tubes are harvested and stabilised using glutaraldehyde. The design provides long-term structural stability of the prosthesis and compliance that is similar to that of an autologous artery. There are no randomised studies comparing the Omniflow II graft to either autologous vein or PTFE. Extensive in vivo testing has been performed for safety and efficacy. The Omniflow graft is registered in Europe, Australia, Canada and in a range of countries in South America and South East Asia.

Methods

All patients between the ages 20 to 90 with peripheral arterial disease with severe, life-style limiting claudication, rest pain or tissue lesions based on occlusion of the femoral or popliteal artery can be considered, if no suitable vein is available for the reconstruction in infrapopliteal reconstructions. Written consent is obtained from all volunteering patients including willingness to participate in the follow-up process. Primary end point of the study is primary patency, defined by duplex scan as freedom from binary restenosis of 50%.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 to 90
* Peripheral arterial occlusive disease with life-style limitation, claudication, rest pain, tissue loss,
* No suitable vein for reconstruction available
* Written consent obtained

Exclusion Criteria

* Acute limb threatening ischaemia
* Patient younger than 20
* Pregnant women
* Myocardial infarction during past 30 days
* Stroke
* Life expectancy < 1 year

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
primary patency, defined by duplex scan as freedom from binary restenosis of 50% | 36 months

SECONDARY OUTCOMES:
secondary patency | 3 months
limb salvage | 6 months
mortality | 12 months
infections | 18 months
reinterventions | 24 and 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Jürg Schmiedli, MD, Principal Investigator — Bern University Hospital
Locations (1):
- Dept. of Cardiovascular Surgery, Bern, Switzerland

REFERENCES:
- [Background] Schmidli J, Savolainen H, Heller G, Widmer MK, Then-Schlagau U, Baumgartner I, Carrel TP. Bovine mesenteric vein graft (ProCol) in critical limb ischaemia with tissue loss and infection. Eur J Vasc Endovasc Surg. 2004 Mar;27(3):251-3. doi: 10.1016/j.ejvs.2003.12.001. PMID 14760592
- [Background] Miller JH, Foreman RK, Ferguson L, Faris I. Interposition vein cuff for anastomosis of prosthesis to small artery. Aust N Z J Surg. 1984 Jun;54(3):283-5. doi: 10.1111/j.1445-2197.1984.tb05318.x. PMID 6380479
- [Background] Kal'noi MP, Mikhailichenko IuP, Alabovskii IuI, Mishin FI. [Experience in medical service to the population in mass agricultural operations in Ipatovo District]. Zdravookhr Ross Fed. 1979;(7):10-3. No abstract available. Russian. PMID 157650
- [Background] Walluscheck KP, Bierkandt S, Brandt M, Cremer J. Infrainguinal ePTFE vascular graft with bioactive surface heparin bonding. First clinical results. J Cardiovasc Surg (Torino). 2005 Aug;46(4):425-30. PMID 16160689
- [Background] Kersting S, Ockert D, Zimmermann T, Meichelbock W, Saeger HD, Bergert H. Infragenicular polytetrafluoroethylene bypass with tapered versus straight vascular grafts: results from a prospective multicenter cohort study. Ann Vasc Surg. 2004 Jul;18(4):440-7. doi: 10.1007/s10016-004-0052-3. PMID 15164262
- [Background] Panneton JM, Hollier LH, Hofer JM. Multicenter randomized prospective trial comparing a pre-cuffed polytetrafluoroethylene graft to a vein cuffed polytetrafluoroethylene graft for infragenicular arterial bypass. Ann Vasc Surg. 2004 Mar;18(2):199-206. doi: 10.1007/s10016-004-0012-y. PMID 15253256
- [Background] Jensen LP, Lepantalo M, Fossdal JE, Roder OC, Jensen BS, Madsen MS, Grenager O, Fasting H, Myhre HO, Baekgaard N, Nielsen OM, Helgstrand U, Schroeder TV. Dacron or PTFE for above-knee femoropopliteal bypass. a multicenter randomised study. Eur J Vasc Endovasc Surg. 2007 Jul;34(1):44-9. doi: 10.1016/j.ejvs.2007.01.016. Epub 2007 Apr 2. PMID 17400486
- [Background] Koch G, Gutschi S, Pascher O, Fruhwirth H, Glanzer H. Analysis of 274 Omniflow Vascular Prostheses implanted over an eight-year period. Aust N Z J Surg. 1997 Sep;67(9):637-9. doi: 10.1111/j.1445-2197.1997.tb04614.x. PMID 9322703
- [Background] Diehm N, Baumgartner I, Jaff M, Do DD, Minar E, Schmidli J, Diehm C, Biamino G, Vermassen F, Scheinert D, van Sambeek MR, Schillinger M. A call for uniform reporting standards in studies assessing endovascular treatment for chronic ischaemia of lower limb arteries. Eur Heart J. 2007 Apr;28(7):798-805. doi: 10.1093/eurheartj/ehl545. Epub 2007 Feb 22. PMID 17317699